CLINICAL TRIAL: NCT05390437
Title: Nutritional Intervention For The Treatment Of Uncomplicated Severe Acute Malnutrition in South Punjab Pakistan
Brief Title: Nutritional Intervention For The Treatment Of Uncomplicated SAM
Acronym: SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanaullah Iqbal (Other)
Collaborators: University of the Punjab (Other)
Responsible Party: Sponsor-Investigator, Sanaullah Iqbal, Associate Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Organization: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Uncomplicated SAM
Record Dates: First submitted 2021-12-13; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Child Nutrition Disorders
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): starch (placebo) 4 grams per day for 60 days
  Interventions: Dietary Supplement: Ready to use theraputic food (RUTF) and Starch (placebo)
- Interventional group (Experimental): Prebiotics (GOS) Galactooligosaccharides 4 gram per day for 60 days
  Interventions: Dietary Supplement: Nutritional intervention with Ready to use theraputic food (RUTF) and prebiotic GOS (galacto oligosaccharides) in combination

INTERVENTIONS:
Dietary Supplement: Nutritional intervention with Ready to use theraputic food (RUTF) and prebiotic GOS (galacto oligosaccharides) in combination — 4gm of prebiotic GOS ( Galactooligosaccharides) and Ready to use theraputic food (RUTF) as per WHO standard on daily basis for 60 Days
  Arms: Interventional group
Dietary Supplement: Ready to use theraputic food (RUTF) and Starch (placebo) — Ready to use therapeutic food (RUTF) as per WHO standard and (Starch Placebo) soluble in water and mix in food on daily basis for 60 Days
  Arms: control group

SUMMARY:
nutritional intervention with ready to use therapeutic food (plumpy nut. by Unicef) and Prebiotics supplimentation ( Galactooligosaccarides). will be given to uncomplicated severe acute malnourished children of 06 months to 59 months of age in southern Punjab Pakistan.one group will be given Ready to use therapeutic food and placebo the other group will be given Prebiotics supplementation (Galacto oligosaccharides) with RUTF ( Ready to use therapeutic Foods).for 60 days primary out will be Mid Upper Arm Circumference >11.5 centimetre

DETAILED DESCRIPTION:
it will be a double blind Randomised Controlled trial in Out Therapeutic Program centres of Teaching Hospital of Dera Ghazi Khan Pakistan children age of 06 months to 59 months of age from the community will be screened out at health centres . Uncomplicated SAM children will be enrolled for study Before intervention there blood sample and stool sample will be sent to the labs for complete blood examination and complete stool examination.

controlled groups will be given Ready To use Therapeutic Food and Placebo (starch) 4 grams per day for 60 days Intervention group will be given Ready to use Therapeutic Food and Prebiotic ( Galactoligosaccharides 4 gram per day for 60 days

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated Severely Acute Malnourished Children

Exclusion Criteria:

* Severely Acute Malnourished children with complication

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Nutritional cure | 60 Days
  Mid Upper Arm Circumference of left arm is measured at the mid point between the tips of shoulder and elbow.It is measured by MUAC tape . More than 11.5 centimetre according to WHO criteria will be primary outcome

SECONDARY OUTCOMES:
Weight gain in kilograms | 60 Days
  weight will be measured on electronic scale on a flat level surface

CONTACTS AND LOCATIONS:
Overall Officials: javeria saleem, pub. health, Principal Investigator — University of Punjab
Locations (1):
- DG Khan, Dera Ghazi Khan, Punjab Province, Pakistan